CLINICAL TRIAL: NCT00830973
Title: Tamoxifen Pharmacogenomics and the Prevention of Recurrent Breast Cancer
Brief Title: The Clinical and Economic Impact of Pharmacogenomic Testing for Tamoxifen Metabolism in Postmenopausal Women Receiving Tamoxifen for Prevention of Recurrent Breast Cancer
Acronym: MHSLabCorp1
Status: Completed | Type: Observational
Sponsor: Medco Health Solutions, Inc. (Industry)
Collaborators: Laboratory Corporation of America (Industry); International Business Machines (IBM) (Industry); Indiana University School of Medicine (Other); Mayo Clinic (Other)
Responsible Party: Robert Epstein, MD, MS, Medco Health Solutions, Inc.
Other Study IDs: MedcoTamoxifen1
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Breast Neoplasms; Tamoxifen
Keywords: Estrogen Antagonists; Antineoplastic Agents, Hormonal; Hormone Antagonists; Hormones; Hormone Substitutes; Selective Estrogen Receptor Modulators; Estrogen Receptor Modulators; Neoplasms; Neoplasms by Site
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasms by Site

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swab
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Active Study Group: The active study group consists of 50 year or older postmenopausal women taking tamoxifen for the prevention of reoccurrence of breast cancer, do not meet exclusion criteria, meet all inclusion criteria, and are enrolled members for Medco clients agreeing to participate.
  Interventions: Other: Poor Metabolism Status Follow Up Therapy Considerations; Other: CYP2D6 Inhibiting Drugs

INTERVENTIONS:
Other: Poor Metabolism Status Follow Up Therapy Considerations — If the patient's CYP2D6 metabolism status is 'poor' then specialist pharmacist will discuss drug therapy alternatives to tamoxifen.
  Other Names: Poor Metabolism
Other: CYP2D6 Inhibiting Drugs — If the patient after having a CYP2D6 test has any drugs that inhibit tamoxifen metabolism then specialist pharmacist will contact the physician for alternative drug therapies.

SUMMARY:
This study will assess the impact of CYP450 2D6 genotype pharmacogenetic testing and the corresponding prescribing impact for postmenopausal women using tamoxifen in a patient care setting for prevention of recurrent breast cancer.

DETAILED DESCRIPTION:
Tamoxifen is a non-steroidal hormonal drug with weak estrogen agonist and potent estrogen antagonist actions. The liver CYP450 metabolic enzyme systems are responsible for metabolizing tamoxifen (the pro-drug form) into its active metabolites. A secondary tamoxifen metabolite known specifically as 4-hydroxy-N-desmethyl-tamoxifen or endoxifen is recognized as the principal potent metabolite responsible for tamoxifen suppression of estrogen-dependent cell proliferation, the stimulus for breast tumor growth. Biotransformation to endoxifen is through the CYPP450 2D6 pathway; therefore, the ability of tamoxifen to effectively suppress breast cancer is jeopardized in patients with certain CYP450 2D6 genetic variants and/or those receiving drug therapy that are known to alter CYP450 2D6 function (i.e., with CYP450 2D6 inhibitors).

Four phenotype expressions classified as ultrarapid, extensive, intermediate and poor metabolizers can be discerned from genotype testing for CYP450 2D6 activity. Patients with normal metabolic activity are known as extensive metabolizers given that they possess either two (genotype = wt/wt) or one (genotype = wt/vt) functioning CYP450 2D6 gene that converts a sufficient amount of tamoxifen in to its active form. Intermediate metabolizers have at least some or very low CYP450 2D6 activity and there does not appear to be uniform consensus on the impact of this phenotype on tamoxifen drug disposition. Poor metabolizers lack any functional CYP450 2D6 activity, and therefore, they do not metabolize tamoxifen enough to produce sufficient endoxifen activity. Approximately 10% of patients (7% of Caucasians and 1-3% of other ethnic groups) are poor metabolizers with a complete absence of CYP450 2D6 activity.

The genetic variants associated with diminished or absent CYP450 2D6 activity are found on CYP450 2D6 alleles *3, *4, *5, *6 and *10. The *3, *4, *5 and *6 alleles, when present in variant form (genotype = vt/vt), account for approximately 97% of nonfunctional CYP450 2D6 variants in caucasians. Of these mutations, those in CYP450 2D6 *4 are most significant for endoxifen.

Poor metabolizer phenotype has been associated with worse relapse-free breast cancer survival and increased risk (up to three times that of intermediate metabolizer status who have some CYP450 2D6 activity) for breast cancer recurrence.

Diagnostic technology now exists to aid in determining which tamoxifen patients are potentially receiving suboptimal treatment from existing alterations in one or more of the approximately 80 alleles of the gene coding for the CPYP450 2D6 enzyme. Recognition of this phenomenon provides physicians and their patients the opportunity for considering the use of other anti-estrogen drugs such as aromatase inhibitors in women whose CYP450 2D6 phenotype puts them at risk for poor response to tamoxifen therapy.

This study will use this diagnostic technology to determine a patient's phenotype provide additional clinical information and alternative drug therapies to the patient's physician.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently has a pharmacy benefit with Medco for an enrolled client
* Patient has a adjudicated tamoxifen pharmacy claims within the last six months
* Patient is still taking tamoxifen to prevent recurrent breast cancer
* Patient is a natural postmenopausal women 50 years of age or older
* Patient signs consent
* Patient is willing to provide sample for genetic testing
* Physician managing tamoxifen therapy is willing to order pharmacogenetic test

Exclusion Criteria:

* Patient is male
* Patient is under 50 years old
* Patient has previous history of CYP450 2D6 testing
* Patient is no longer taking tamoxifen
* Patient refuses to sign consent
* Patient wishes to no longer participate after testing
* Patient's physician refuses to order pharmacogenetic test

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The active study group consists of 50 year or older postmenopausal women taking tamoxifen for the prevention of reoccurrence of breast cancer, do not meet exclusion criteria, meet all inclusion criteria, and are enrolled members for Medco clients agreeing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of different CYP450 2D6 phenotypes including poor metabolism status | 14 months

SECONDARY OUTCOMES:
Determine the prevalence of concomitant drug therapy involving tamoxifen and potent CYP450 2D6 inhibitors | 14 months
Determine the effect of CYP450 2D6 genotyping that indicates poor metabolism status has on physician willingness to change tamoxifen therapy within 60 days of receiving test results and accompanying interpretations | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Epstein, MD, MS, Principal Investigator — Medco Health Solutions, Inc.
Locations (1):
- Robert Epstein, Franklin Lakes, New Jersey, United States